CLINICAL TRIAL: NCT07103187
Title: The Role of Prebent Titanium Mesh With 3D-Printed Model in Reconstruction of Zygomatico-Orbital Fractures
Brief Title: Evaluating The Prebent Titanium Mesh for Zygomatico-Orbital Reconstruction in Twelve Patients Measuring Multiple Ophthalmologic Parameters, Aesthetic Results, Orbital Volume, Area of Bone Defect, Layout Angle, Gab Length and The Accuracy of Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, AYMAN M. ARAKEEP, MSc, PhD researcher, Assistant Lecturer of Oral & Maxillofacial Surgery, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-OS-1-19-8
Record Dates: First submitted 2025-07-28; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Zygomaticomaxillary Complex Fracture; Orbital Floor Fractures; Ophthalmic Trauma
Keywords: Orbital reconstruction; Orbital fractures; Automatic segmentation; 3D orbital analysis; Orbital volume; Orbito-zygomatico-maxillary complex fracture
MeSH Terms: conditions — Orbital Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Only single arm of the study (Experimental): This is the only arm of the study containing 12 patients who will be operated for reconstruction for unilateral OZMC fracture. A lot of outcome measures will be measured to evaluate the effectiveness of the intervention.
  Interventions: Procedure: Zygomatico-Orbital reconstruction

INTERVENTIONS:
Procedure: Zygomatico-Orbital reconstruction — Zygomatico-Orbital reconstruction was done by ORIF for the zygomatic complex fractures at multiple suture lines by mini plates and screws. Orbital floor reconstruction was done mainly by using a prebent titanium mesh on a 3D printed model.

SUMMARY:
Purpose: The aim of this study was to evaluate the role of using a prebent titanium mesh on a 3D-printed model as an intraoperative guide to reconstruct orbito-zygomatic-maxillary complex (OZMC) fractures.

Subjects and method: This is a prospective, interventional, longitudinal, single armed case series study that was carried out on twelve patients with unilateral displaced orbito-zygomatico-maxillary complex (OZMC) fracture indicated for orbital floor reconstruction as evidenced by clinical and radiographic examination. Open reduction and internal fixation were utilized to treat those fractures, patients were collected from the department of Oral and Maxillofacial surgery, Faculty of Dentistry, Tanta University. Post-operative evaluation: all patients underwent regular follow up for six months. The following parameters were evaluated: visual acuity, external appearance of the eye including hypoglobus and enophthalmos, diplopia, ocular motility, the aesthetic results, orbital volume, area of bone defect, layout angle, gab length and the zygomatic reconstruction.

DETAILED DESCRIPTION:
This study was conducted on twelve patients with unilateral displaced OZMC fracture indicated for orbital floor reconstruction as evidenced by clinical and radiographic examination. The patients' ages ranged from 18-55 years old. All patients were evaluated preoperatively for collecting demographic data, taking general medical, surgical, and dental history and for determining the main patient's chief complaints and postoperative expectations. Approval for this project was obtained from Research Ethics Committee (REC) of faculty of Dentistry, Tanta University. The purpose of the present study was explained to the patients and informed consents were obtained according to the guidelines of human research adopted by the REC at Faculty of Dentistry, Tanta University. After obtaining the preoperative CT scan, 3D simulation was performed using (3Diagnosys, version 4.2, 3diemme. Como, Italy) as the following steps:

1. Importing CT DICOM images.
2. Mirror image of the normal side.
3. Segmentation to remove any unwanted areas.
4. Thresholding to choose the density of bone.
5. Conversion to STL format.
6. Exporting as an STL file to the 3D printer. The 3D printer (Upbox, Tiertime, Korea) was used to print the patient specific model. The Printing material was ABS/PLA. The technology used for the printing process was FDM (Fused Deposition Modeling), where a filament is heated above 200 degrees and extruded through a nozzle of 0.4 mm diameter to print layer by layer with a resolution of 100 microns. Routine preoperative investigations (complete blood picture, prothrombin test, liver &renal function test and viral profile) were done for all patients, together with relevant medical consultation when required. The patients were operated under general anesthesia via nasal endotracheal intubation. The surgical site was disinfected using Povidone-iodine then isolated and draped with sterile dressing. Reconstruction was done carefully. All outcome measures were measured later on, and adequate statistical analysis was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral displaced zygomatico-orbital fracture (with fractured orbital floor).
2. Patients with no previous history of orbital reconstruction.
3. Diplopia within 30° of primary gaze.
4. Radiological evidence of extraocular muscle entrapment and/or positive forced duction test.
5. Enophthalmos of more than 2mm.

Exclusion Criteria:

1. Bilateral zygomatico-orbital fractures.
2. Rupture of the globe.
3. Hyphema.
4. Retinal detachment.
5. Traumatic optic nerve lesions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Orbital volume | Preoperatively. Postoperatively within two weeks after the operation.
  By obtaining CT scan of the face then the DICOM data was imported by BONELOGIC CMF ORBITAL software provided by Disior company which performed automated 3D analysis for the orbits preoperatively and postoperatively.
Area of bone defect (Orbital symmetry) | Preoperatively. Postoperatively within two weeks after the operation.
  By obtaining CT scan of the face then the DICOM data was imported by BONELOGIC CMF ORBITAL software provided by Disior company which performed automated 3D analysis for the orbits preoperatively and postoperatively.
Acuraccy of Orbito-Zygomatico-maxillary complex fracture reconstruction | Only postoperatively within two weeks after the operation.
  On a postoperative CT scan of the face adequate zygomatic reduction was judged by evaluating any involved parts from the following reference points, including zygomaticofrontal suture, zygomatico-sphenoidal suture, zygomaticomaxillary buttress, inferior orbital rim, and zygomatic arch, which was judged by two experienced surgeons as good, satisfactory or poor.

SECONDARY OUTCOMES:
Visual acuity | Preoperative. Postoperatively 2 weeks, 1 month, 2 months, 3 months and 6 months.
  Measured by distance eye chart.
Vertical dystopia | Preoperative. Postoperatively 2 weeks, 1 month, 2 months, 3 months and 6 months.
  Measured by drawing an imaginary line horizontally across the patient's inter-pupillary axis and determine if the pupil of the affected eye is in the lower level in relation to the intact eye which revealed hypoglobus.
Enophthalmos | Preoperative. Postoperatively 2 weeks, 1 month, 2 months, 3 months and 6 months.
  Measured by the aid of exophthalmometer represented by four grades from 0 to 3 as follows: grade 0 = no enophthalmos, grade 1= mild enophthalmos (less than 1 mm), grade 2= moderate enophthalmos (ranged from 1 to 2 mm), grade 3= severe enophthalmos (over 2mm).
Diplopia | Preoperative. Postoperatively 2 weeks, 1 month, 2 months, 3 months and 6 months.
  Assessed if it was present in the primary position of gaze, within 30° degree or in a secondary position of gaze depending on the patient response by specialized ophthalmologist.
Ocular motility | Preoperative. Postoperatively 2 weeks, 1 month, 2 months, 3 months and 6 months.
  Tested by asking the patient to follow a moving target into the diagnostic positions of gaze observing the extent of movement of each eye. The amount of limitation of movement is classified as grade 1= slight limitation, grade 2= moderate limitation, grade 3= marked limitation or grade 4= no movement according to the observation of two independent examiners.
The layout angle | Only postoperatively within two weeks after the operation.
  Measured on a postoperative CT scan of the face and defined as an acute angle between the titanium mesh and an arbitrary line representing the premorbid status of the orbital floor connecting the starting point of the orbital floor fracture to its end. This line reflects the normal bone contour and is easy to suppose from contralateral normal orbital floor.
The gap length | Only postoperatively within two weeks after the operation.
  Measured on a postoperative CT scan of the face and defined as the distance from the distal tip of the titanium mesh to the posterior bone shelf margin.

OTHER OUTCOMES:
Aesthetic results | 6 months postoperatively.
  Which were judged by means of photographs using the 3-score scale as "good", "satisfactory", and "poor".

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Algharbiah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All patient data without any identity show could be available by request from the corresponding author including clinical photos and raw tables for all data entry of the study
Supporting Information: Study Protocol, ICF
Time Frame: The data could be available after publication within 6 months from now.
Access Criteria: The data will be held on a private cloud and access will be provided upon request from the corresponding author.